CLINICAL TRIAL: NCT04046575
Title: Phase I Study of Radiation Dose Intensification With Accelerated Hypofractionated Intensity Modulated Radiation Therapy and Concurrent Carboplatin and Paclitaxel for Inoperable Esophageal Cancer
Brief Title: Radiation Dose Intensification With Accelerated Hypofractionated Intensity Modulated Radiation Therapy and Concurrent Carboplatin and Paclitaxel for Inoperable Esophageal Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201909019
Record Dates: First submitted 2019-08-02; First posted 2019-08-06 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Esophagus Cancer; Esophageal Cancer; Cancer of the Esophagus
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Carboplatin; Blood Specimen Collection; Circulating Tumor DNA; squamous cell carcinoma-related antigen; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- IMRT + Carboplatin + Paclitaxel (Experimental): Concurrent chemoradiation will consist of hypofractionated intensity modulated radiation therapy (IMRT) with simultaneous integrated boost (SIB) for 3 weeks with carboplatin and paclitaxel for 3 cycles every 7 days. Endoscopy and (optional) PET/CT within 6-8 weeks post-completion of chemoradiation.
  Interventions: Radiation: Intensity Modulated Radiation Therapy; Drug: Carboplatin; Other: MD Anderson Symptom Inventory (MDASI)-Plus module; Other: EuroQol (EQ-5D); Other: SF-12; Other: MOS Social Support Measure; Other: CES-D; Procedure: Blood for ctDNA (optional); Procedure: Blood for SCCA; Drug: Paclitaxel

INTERVENTIONS:
Radiation: Intensity Modulated Radiation Therapy — -15 fractions of treatment
  Other Names: IMRT
Drug: Carboplatin — Begins on day 1 of radiotherapy
  Other Names: Paraplatin
Other: MD Anderson Symptom Inventory (MDASI)-Plus module — The QOL questionnaires will be answered by the patients prior to the start of chemoradiation, on the last week of RT, and at 6-8 week follow-up, 3, 6, 9, and 12 months post completion of RT
Other: EuroQol (EQ-5D) — The QOL questionnaires will be answered by the patients prior to the start of chemoradiation, on the last week of RT, and at 6-8 week follow-up, 3, 6, 9, and 12 months post completion of RT
Other: SF-12 — The QOL questionnaires will be answered by the patients prior to the start of chemoradiation, on the last week of RT, and at 6-8 week follow-up, 3, 6, 9, and 12 months post completion of RT
Other: MOS Social Support Measure — The QOL questionnaires will be answered by the patients prior to the start of chemoradiation, on the last week of RT, and at 6-8 week follow-up, 3, 6, 9, and 12 months post completion of RT
Other: CES-D — The QOL questionnaires will be answered by the patients prior to the start of chemoradiation, on the last week of RT, and at 6-8 week follow-up, 3, 6, 9, and 12 months post completion of RT
Procedure: Blood for ctDNA (optional) — -Collected at pre-treatment, every 2 weeks during chemoradiation, every 2-3 weeks during consolidation chemotherapy, completion of therapy, 6-8 week follow-up, 3 month follow-up, 6 month follow-up, and 12 month follow-up
Procedure: Blood for SCCA — -Collected at pre-treatment, completion of therapy, and 6 month follow-up
Drug: Paclitaxel — Begins on day 1 of radiotherapy
  Other Names: Taxol

SUMMARY:
Rates of local disease control in patients with locally advanced esophageal cancer who are not candidates for surgical resection are suboptimal. Despite treatment with chemotherapy and radiation therapy approximately half of patients will develop recurrence of their cancer at the site of the original primary cancer. Salvage therapy options are largely ineffective and nearly all patients who develop local disease recurrence will succumb to their cancer. Recent clinical trials for lung cancer have demonstrated that local tumor control can be improved safely with accelerated hypofractionated radiation therapy regimens in order to achieve radiation dose intensification. This clinical trial aims to adapt those techniques and assess the safety of such a regimen for the treatment of inoperable thoracic esophageal cancers.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven carcinoma of the thoracic esophagus, or gastroesophageal junction (GEJ).
* Amenable to definitive chemoradiation.
* Unresectable esophageal cancer or not a surgical candidate as determined by a surgeon or multidisciplinary tumor board.
* At least 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Complete blood count (CBC) with differential obtained within 30 days prior to registration with adequate bone marrow function:

  * Absolute neutrophil count (ANC) ≥1,500 cells/mm3
  * Platelets ≥100,000 cells/ mm3
  * Hemoglobin ≥9 g/dL (transfusion or other intervention to achieve hemoglobin ≥9 g/dL is acceptable).
* Adequate renal function within 30 days prior to registration: Serum creatinine ≤ 1.5x upper limit of normal or calculated creatinine clearance ≥ 50 mL/min within 30 days prior to registration estimated by the Cockcroft-Gault formula:

Creatinine Clearance (male) = [(140 - age) x (wt in kg)] [(Serum Creatinine mg/dl) x (72)] Creatinine Clearance (female) = 0.85 x Creatinine Clearance (male)

*Adequate hepatic function within 30 days prior to registration: bilirubin ≤ 1.5x upper limit of normal, ALT/AST ≤3 x upper limit of normal (ULN).

* Negative pregnancy test within 14 days of registration or otherwise be determined to not be of childbearing potential. Postmenopausal women must be amenorrheic for 12 months or more. Women of childbearing potential must agree to perform appropriate contraception methods and not breastfeed until 30 days after last chemotherapy.
* Planned to undergo IMRT with photon beam radiation therapy. 3D CRT and proton modalities are not allowed.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Primary cervical esophageal cancer
* Siewert-Stein Type III carcinomas of the stomach.
* Esophageal perforation, fistula, or deep ulceration to the mediastinum.
* Currently receiving any other investigational agents.
* Known brain metastases. Patients with known brain metastases must be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to carboplatin, paclitaxel, or other agents used in the study.
* Planning to undergo or has already undergone induction chemotherapy.
* Presence of any active malignancy within 2 years that may alter the course of esophageal cancer therapy.
* Prior radiation therapy to the neck, thorax, or abdomen is not allowed UNLESS there is expected to be no overlap with the study esophageal radiotherapy treatment. Prior radiation therapy treatment plan reports must be reviewed by study PI to verify no overlap of treatment fields.
* Severe active comorbidity as defined below:

  * Unstable angina and/or congestive heart failure within the last 6 months.
  * Transmural myocardial infarction within the last 6 months.
  * History of stroke, cerebral vascular accident, or transient ischemic attack within the last 6 months.
  * Serious and inadequately controlled cardiac arrhythmia
  * Bacterial or fungal infection requiring intravenous antibiotics at the time of registration.
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration.
  * Peripheral neuropathy > grade 1 at time of registration.
* Persistent complications from any major surgery within 4 weeks of study treatment start.
* Any other major medical illness that in the investigator's opinion would prevent safe administration or completion of protocol therapy.
* Pregnant or lactating woman. Women of childbearing potential with positive pregnancy test at baseline, or women who have not taken a pregnancy test at baseline. A man or woman who does not agree to use appropriate contraception.
* Patients with HIV are eligible unless their CD4+ T-cell counts are < 350 cells/mcL or they have a history of AIDS-defining opportunistic infection within the 12 months prior to registration. Concurrent treatment with effective ART according to DHHS treatment guidelines is recommended.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2029-11-20 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of hypofractionated IMRT with chemotherapy | Through 6 month follow-up for all enrolled patients (estimated to be 65 months)
  The MTD of the combination of radiation and FOLFOX will be estimated using the proposed TITE-CRM model. After the phase I study, the MTD will be chosen as the dose that yields a posterior toxicity estimate closest to 20% while being between 15% and 25%. Toxicity will be coded using CTCAE v5.0.

SECONDARY OUTCOMES:
Median local relapse-free survival | Through completion of follow-up (up to 6 years)
  -The length of time after treatment ends that the participants survives without any signs or symptoms of the cancer recurring within the radiated field
Median overall survival | Through completion of follow-up (up to 6 years)
  -The length of time from the start of treatment that participants are still alive
Median progression-free survival | Through completion of follow-up (up to 6 years)
  -The length of time from the start of treatment to progression or death from any cause
Patient reported outcomes as measured by the MDASI-Plus | From baseline through 12 months post end of treatment
  * The MDASI-plus is a reliable, validated tool for assessing cancer-related symptoms regardless of therapy or specific cancer diagnosis. Patients are asked to fill out a twenty-seven question inventory, ranking their symptoms on a 0 (no problems) to 10 (worst imaginable) scale
  * The mean of the scores will be calculated at each time point and compared to other time points to assess changes in cancer-related symptoms
Patient reported outcomes as measured by the EQ-5D | From baseline through 12 months post end of treatment
  * standardized 2-part, patient-administered instrument used for direct and indirect assessment of health state utilities
  * The first part asks respondents to "check the ONE box [next to the appropriate statement] that best describes your health TODAY" for each of 5 health dimensions, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The second part of the EQ-5D is a visual analogue scale (VAS) valuing current health state
  * Both the 5-item index score and the VAS score are transformed into a utility score between 0 "Worst health state" and 1 "Best health state
Patient reported outcomes as measured by the SF-12 | From baseline through 12 months post end of treatment
  * 12-item questionnaire measuring physical and mental functional status
  * Mental and physical component scores will be calculated in addition to calculating the measure's eight individual subscales (physical functioning, social functioning, role limitations due to physical problems, body pain, general health, role limitations due to emotional problems general health, vitality, and mental health). Higher scores indicate better quality of life
Patient reported outcomes as measured by the MOS Social Support | From baseline through 12 months post end of treatment
  -19 items
  -. Response choices range from "none of the time" (1) to "all of the time" (5). A mean social support score for all 19 items is computed with higher scores indicating a greater availability of social support.
Patient reported outcomes as measured by the 4-Item CES-D | From baseline through 12 months post end of treatment
  * 4 item screening version to evaluate depressive symptoms
  * The mean of the scores will be calculated at each time point and compared to other time points to assess changes in depression symptoms
Number and type of adverse events experienced by patient | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Vlacich, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu